CLINICAL TRIAL: NCT02321046
Title: An epidemiOlogy Study to deteRmine the Prevalence of EGFR muTations in RUSsian Patients With Advanced NSCLC (ORTUS)
Brief Title: An epidemiOlogy Study to deteRmine the Prevalence of EGFR (Epidermal Growth Factor Receptor) muTations in RUSsian Patients With Advanced NSCLC (Non-Small Cell Lung Cancer).
Acronym: ORTUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00101
Record Dates: First submitted 2014-11-27; First posted 2014-12-22 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer, NSCLC, Epidermal growth factor receptor, EGFR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cytology and plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multicentre, non-interventional, prospective study to be carried out in representative oncology departments / institutions in order to determine the prevalence of EGFR mutations in treatment-naive Russian patients with cytologically verified advanced NSCLC in Russia.

DETAILED DESCRIPTION:
This is a multicentre, non-interventional, prospective study to be carried out in representative oncology departments / institutions in order to determine the prevalence of EGFR mutations in treatment-naive Russian patients with cytologically verified advanced NSCLC in Russia. No additional procedures besides those already used in the routine clinical practice will be applied to the patients. Treatment assignment will be done according to the current practice.

It is planned to enrol approximately 300 subjects in Russian Federation. Approximately 60 EGFR m+ (mutation-positive) patients will be followed for 1.5 years.

EGFR mutations rate before treatment in cytology and plasma samples in treatment-naive patients with advanced NSCLC in Russia is considered as the primary outcome variable in this study.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically verified advanced (stages IIIB - IV) nonsquamous (adenocarcinoma, large cell carcinoma) and mixed subtypes of NSCLC and NSCLC-NOS), diagnosed before enrolment into the study
* Quality and quantity of the cytological sample material meeting the requirements of the molecular-genetic testing
* No previous/ ongoing treatment for NSCLC at the moment of recruitment

Exclusion Criteria:

* Squamous NSCLC cytologically confirmed subtype of cancer
* Any medical condition which on the opinion of the investigator may interfere the patient's participation in the study
* Quality and quantity of the cytological sample material insufficient for the molecular-genetic testing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Target study population will be treatment-naive patients of both sexes, 18 years and older, with cytologically-verified advanced (stage IIIB-IV) non-squamous, mixed subtypes of NSCLC and NSCLC-NOS (Non-Small Cell Lung Cancer - Not Otherwise Specified), diagnosed before enrolment into the study, consented to participate in this non-interventional study, who visit the oncology hospitals/departments in the Russian Federation.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
EGFR mutations (EGFR del746-750, EGFR L858R, EGFR T790M) rate in cytology and plasma samples prior to treatment | up to 18 months

SECONDARY OUTCOMES:
Patient characteristics: Gender. Age. Race, ethnicity. Smoking habits. Family history of NSCLC. | up to 18 months
Disease information/diagnostic procedures | up to 18 months
  Date of the cytological verification of the NSCLC diagnosis. Disease stage and TNM classification. Morphological classification. Extent of the disease. Performance Status ECOG, including at diagnosis
EGFR mutations profile in cytology and/or histology (depending on the availablility of samples) and plasma samples at the time of every progression or in 1.5 year follow up in case of no progression | up to 18 months
Characteristics of the 1st line and subsequent lines of antitumor therapy | up to 18 months
  1st line and subsequent lines of therapy treatment, therapy regimen, medicines used for therapy (drugs by INN), for EGFRm+ patients - number of cycles of antitumor therapy, onset date, end date of each line
Clinical outcome/Patient response (for EGFRm+ patients who entered observation phase) | up to 18 months
  Treatment response/ progression of disease on every line of antitumor therapy: progressive disease, partial response, stable disease and complete response according to RECIST 1.1 evaluation and/or any other clinical assessment.
  Death: Disease-related or for other reasons

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bedenkov, MCMD, Study Director — AstraZeneca; Konstantin Lactionov, Professor, Principal Investigator — Russian Cancer Research Center named after N.N.Blokhin; Irina Demidova, PHD, Principal Investigator — Moscow City Clinical Cancer Hospital #62
Locations (26):
- Russia (26):
  - Research Site, Khanti-Manskiysk, Russia
  - Research Site, Novisibirsk, Russia
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Chelyabinsk
  - Research Site, Irkutsk
  - Research Site, Kemerovo
  - Research Site, Khabarovsk
  - Research Site, Kirov
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Orenburg
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Tambov
  - Research Site, Tomsk
  - Research Site, Ufa
  - Research Site, Vladivostok
  - Research Site, Volgograd
  - Research Site, Yuzhno-Sakhalinsk

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133FR00101&attachmentIdentifier=50891de4-4c60-4820-a706-750278dc9ea0&fileName=NIS_ORTUS_CSR-Synopsis.pdf&versionIdentifier=